CLINICAL TRIAL: NCT03311724
Title: A Phase 2, Double-Blind, Placebo-Controlled, 3-Month Trial of LY3298176 Versus Placebo in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of Tirzepatide (LY3298176) in Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16860; I8F-MC-GPGF (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Results first posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 4,8,12mg Tirzepatide (Experimental): Participants received Tirzepatide by subcutaneous (SC) injection in three dose escalations starting with 4 milligrams (mg) for four weeks followed by 8mg for four weeks followed by 12mg for four weeks.
  Interventions: Drug: Tirzepatide
- 2.5,5,10,15mg Tirzepatide (Experimental): Participants received Tirzepatide by SC injection in four dose escalations starting with 2.5mg for two weeks followed by 5mg for two weeks followed by 10mg for four weeks followed by 15mg for four weeks.
  Interventions: Drug: Tirzepatide
- 2.5,7.5,15mg Tirzepatide (Experimental): Participants received Tirzepatide by SC injection in three dose escalations starting with 2.5mg for four weeks followed by 7.5mg for four weeks followed by 15mg for four weeks.
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Placebo administered by SC injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: 2.5,5,10,15mg Tirzepatide; 2.5,7.5,15mg Tirzepatide; 4,8,12mg Tirzepatide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy of tirzepatide in participants with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes (T2DM) for ≥6 months according to the Criteria for Diagnosing Type 2 Diabetes Mellitus (American Diabetes Association 2017).
* Have HbA1c of 7.0% to 10.5%, inclusive, as assessed by the central laboratory.
* If on metformin, have been treated with stable doses of metformin for at least 3 months.
* Have a body mass index (BMI) between 23 and 45 (Inclusive) kilograms per square meter.

Exclusion Criteria:

* Have type 1 diabetes (T1D).
* Have used any glucose-lowering medication other than metformin within 3 months prior to study entry or during screening/lead-in period or have used any glucagon-like peptide-1 receptor agonists (GLP-1 RAs) at any time in the past 12 months.
* Have had any of the following cardiovascular conditions: acute myocardial infarction (MI), New York Heart Association Class III or Class IV heart failure, or cerebrovascular accident (stroke).
* Have acute or chronic hepatitis, signs and symptoms of any other liver disease other than nonalcoholic fatty liver disease (NAFLD), or alanine aminotransferase (ALT) level >2.5 times the upper limit of the reference range, as determined by the central laboratory at study entry; participants with NAFLD are eligible for participation in this trial.
* Have had chronic or acute pancreatitis any time prior to study entry.
* Have an estimated glomerular filtration rate (eGFR) <45 milliliters/minute/1.73 square meter, calculated by the Chronic Kidney Disease-Epidemiology (CKD-EPI) equation.
* Have serum calcitonin ≥20 picograms per milliliter, as determined by the central laboratory at study entry.
* Have any condition that is a contraindication for use of the GLP-1 RA class (per country-specific labels) at study entry or develop such condition between study entry and randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- United States (13):
  - Valley Research, Fresno, California
  - National Research Institute, Los Angeles, California
  - Catalina Research Institute, LLC, Montclair, California
  - University Clinical Investigators, Inc., Tustin, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Suncoast Research Group, LLC, Miami, Florida
  - Solaris Clinical Research, Meridian, Idaho
  - Cotton O'Neil Diabetes and Endocrinology Center, Topeka, Kansas
  - Clinical Research Professionals, St Louis, Missouri
  - Aventiv Research, Columbus, Ohio
  - New Phase Research & Development, Knoxville, Tennessee
  - Dallas Diabetes Endocrine Center, Dallas, Texas
  - Consano Clinical Research, Shavano Park, Texas

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Tirzepatide in Participants With Type 2 Diabetes — https://www.lillytrialguide.com/en-US/studies/type-2-diabetes/GPGF#?postal=

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received Placebo by subcutaneous (SC) injection.
- 4, 8 and 12mg Tirzepatide: Participants received Tirzepatide by SC injection in three dose escalations starting with 4mg for four weeks followed by 8mg for four weeks followed by 12mg for four weeks.
- 2.5, 5, 10, and 15mg Tirzepatide: Participants received Tirzepatide by SC injection in four dose escalations starting with 2.5mg for two weeks followed by 5mg for two weeks followed by 10mg for four weeks followed by 15mg for four weeks.
- 2.5, 7.5 and 15mg Tirzepatide: Participants received Tirzepatide by SC injection in three dose escalations starting with 2.5mg for four weeks followed by 7.5mg for four weeks followed by 15mg for four weeks.
Period: Overall Study
Arm/Group | Placebo | 4, 8 and 12mg Tirzepatide | 2.5, 5, 10, and 15mg Tirzepatide | 2.5, 7.5 and 15mg Tirzepatide
Started | 26 | 29 | 28 | 28
Received At Least One Dose of Study Drug | 26 | 29 | 28 | 28
Completed Treatment | 20 | 27 | 22 | 26
Completed | 23 | 28 | 26 | 27
Not Completed | 3 | 1 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 4, 8 and 12mg Tirzepatide | 2.5, 5, 10, and 15mg Tirzepatide | 2.5, 7.5 and 15mg Tirzepatide | Total
Number analyzed (Participants) | 26 | 29 | 28 | 28 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (10.13) | 61.2 (7.56) | 55.5 (8.54) | 56.6 (9.21) | 57.4 (9.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 12 | 5 | 45
  Male | 12 | 15 | 16 | 23 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 15 | 14 | 14 | 59
  Not Hispanic or Latino | 10 | 14 | 14 | 14 | 52
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 1 | 0 | 3
  Asian | 0 | 1 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 7 | 5 | 2 | 15
  White | 25 | 19 | 20 | 23 | 87
  More than one race | 0 | 0 | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 29 | 28 | 28 | 111
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1C] | 8.23 (1.22) | 8.35 (0.897) | 8.48 (1.171) | 8.35 (1.12) | 8.35 (1.094)
Fasting Blood Glucose (FBG) [Mean (Standard Deviation); unit: millimoles per liter (mmol/L)] | 9.68 (3.44) | 9.76 (3.03) | 10.40 (4.04) | 10.67 (4.22) | 10.13 (3.69)
Body Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 89.58 (23.69) | 87.98 (17.35) | 88.74 (18.21) | 89.59 (16.91) | 88.95 (18.87)
Waist Circumference [Mean (Standard Deviation); unit: centimeter (cm)] | 109.09 (15.38) | 107.65 (12.22) | 107.02 (12.64) | 105.10 (12.19) | 107.19 (13.02)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Haemoglobin A1c (HbA1c)
Description: Least squares (LS) mean was calculated using mixed model repeated measures model (MMRM) with baseline + baseline BMI group + baseline metformin flag + treatment + time + treatment*time as fixed factors.
Time Frame: Baseline, 3 Months
Population: All participants who received at least 1 dose of study drug and had baseline and at least one post baseline data. Participants who discontinued study drug or initiated rescue drug were excluded.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1C
Groups:
- Placebo: Placebo administered SC.
Arm/Group | Placebo | 4, 8 and 12mg Tirzepatide | 2.5, 5, 10, and 15mg Tirzepatide | 2.5, 7.5 and 15mg Tirzepatide
Number analyzed (Participants) | 20 | 27 | 23 | 26
Percentage of HbA1C | 0.2 (0.21) | -1.7 (0.19) | -2.0 (0.20) | -1.8 (0.19)
Statistical Analysis 1: Comparison: Placebo vs 4, 8 and 12mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-2.5 to -1.4]
Statistical Analysis 2: Comparison: Placebo vs 2.5, 5, 10, and 15mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-2.8 to -1.7]
Statistical Analysis 3: Comparison: Placebo vs 2.5, 7.5 and 15mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-2.5 to -1.4]

2. Secondary Outcome: Percentage of Participants Achieving HbA1c Target of <7.0%
Description: Percentage of participants achieving HbA1c target of < (less than) 7.0%.
Time Frame: 3 Months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 4, 8 and 12mg Tirzepatide | 2.5, 5, 10, and 15mg Tirzepatide | 2.5, 7.5 and 15mg Tirzepatide
Number analyzed (Participants) | 20 | 27 | 23 | 26
percentage of participants | 10 | 74.1 | 87 | 84.6
Statistical Analysis 1: Comparison: Placebo vs 4, 8 and 12mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 56.54, 95% CI 2-sided [9.43 to 338.97]
Statistical Analysis 2: Comparison: Placebo vs 2.5, 5, 10, and 15mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 183.48, 95% CI 2-sided [22.0 to 999] — Maximum confidential interval is ">999"
Statistical Analysis 3: Comparison: Placebo vs 2.5, 7.5 and 15mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 157.54, 95% CI 2-sided [21.63 to 999] — Maximum confidential interval is ">999"

3. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (FBG)
Description: LSMean was calculated using MMRM model with baseline + baseline HbA1C group + baseline BMI group + baseline Metformin flag + treatment + time + treatment*time as fixed factors.
Time Frame: Baseline, 3 Months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | Placebo | 4, 8 and 12mg Tirzepatide | 2.5, 5, 10, and 15mg Tirzepatide | 2.5, 7.5 and 15mg Tirzepatide
Number analyzed (Participants) | 20 | 27 | 23 | 25
milligrams per deciliter (mg/dL) | -12.3 (9.27) | -60.7 (8.21) | -70.2 (8.72) | -74.2 (8.67)
Statistical Analysis 1: Comparison: Placebo vs 4, 8 and 12mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -48.5, 95% CI 2-sided [-70.6 to -26.3]
Statistical Analysis 2: Comparison: Placebo vs 2.5, 5, 10, and 15mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -58.0, 95% CI 2-sided [-80.7 to -35.2]
Statistical Analysis 3: Comparison: Placebo vs 2.5, 7.5 and 15mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -61.9, 95% CI 2-sided [-84.6 to -39.2]

4. Secondary Outcome: Change From Baseline in Body Weight
Description: as for outcome 3
Time Frame: Baseline, 3 Months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | Placebo | 4, 8 and 12mg Tirzepatide | 2.5, 5, 10, and 15mg Tirzepatide | 2.5, 7.5 and 15mg Tirzepatide
Number analyzed (Participants) | 20 | 27 | 23 | 26
kilogram (kg) | -0.5 (0.86) | -5.3 (0.78) | -5.5 (0.80) | -5.7 (0.79)
Statistical Analysis 1: Comparison: Placebo vs 4, 8 and 12mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -4.8, 95% CI 2-sided [-7.1 to -2.6]
Statistical Analysis 2: Comparison: Placebo vs 2.5, 5, 10, and 15mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -5.0, 95% CI 2-sided [-7.2 to -2.7]
Statistical Analysis 3: Comparison: Placebo vs 2.5, 7.5 and 15mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -5.2, 95% CI 2-sided [-7.5 to -2.9]

5. Secondary Outcome: Change From Baseline in Waist Circumference
Description: as for outcome 3
Time Frame: Baseline, 3 Months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: centimeter (cm)
Arm/Group | Placebo | 4, 8 and 12mg Tirzepatide | 2.5, 5, 10, and 15mg Tirzepatide | 2.5, 7.5 and 15mg Tirzepatide
Number analyzed (Participants) | 20 | 27 | 23 | 26
centimeter (cm) | -2.5 (1.01) | -4.8 (0.90) | -4.9 (0.94) | -4.9 (0.93)
Statistical Analysis 1: Comparison: Placebo vs 4, 8 and 12mg Tirzepatide; Test type: Superiority; p = 0.075, Mixed Models Analysis; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-4.7 to 0.2]
Statistical Analysis 2: Comparison: Placebo vs 2.5, 5, 10, and 15mg Tirzepatide; Test type: Superiority; p = 0.065, Mixed Models Analysis; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-4.9 to 0.1]
Statistical Analysis 3: Comparison: Placebo vs 2.5, 7.5 and 15mg Tirzepatide; Test type: Superiority; p = 0.065, Mixed Models Analysis; Mean Difference (Final Values) = -2.4, 95% CI 2-sided [-4.9 to 0.2]

6. Secondary Outcome: Number of Participants With Anti Drug Antibodies
Description: Number of participants with anti drug antibodies.
Time Frame: Baseline through 3 Months
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | 4, 8 and 12mg Tirzepatide | 2.5, 5, 10, and 15mg Tirzepatide | 2.5, 7.5 and 15mg Tirzepatide
Number analyzed (Participants) | 25 | 29 | 28 | 27
participants | 0 | 10 | 8 | 4

7. Secondary Outcome: Number of Episodes of Total Hypoglycemia Episodes
Description: Number of episodes of total hypoglycemia episodes with plasma glucose <= ( less than or equal to) 54 mg/dL.
Time Frame: Baseline through 3 Months
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: Episodes
Arm/Group | Placebo | 4, 8 and 12mg Tirzepatide | 2.5, 5, 10, and 15mg Tirzepatide | 2.5, 7.5 and 15mg Tirzepatide
Number analyzed (Participants) | 26 | 29 | 28 | 28
Episodes | 0 | 0 | 0 | 1

8. Secondary Outcome: Pharmacokinetics (PK): Average Trough Concentration (Conctrough) of Tirzepatide
Description: Pharmacokinetics (PK): Average Trough Concentration (Conctrough) of Tirzepatide.
Time Frame: Week 4, 8 12: Pre-dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK samples.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 4, 8 and 12mg Tirzepatide | 2.5, 5, 10, and 15mg Tirzepatide | 2.5, 7.5 and 15mg Tirzepatide
Number analyzed (Participants) | 29 | 28 | 28
nanograms per milliliter (ng/mL) | 508 (366) | 704 (518) | 630 (414)

ADVERSE EVENTS:
Time Frame: Baseline through end of study (Up to 15 weeks).
Description: All randomized participants.
Arm/Group | Placebo | 4, 8 and 12mg Tirzepatide | 2.5, 5, 10, and 15mg Tirzepatide | 2.5, 7.5 and 15mg Tirzepatide
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/29 | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/26 | 1/29 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 7/26 | 19/29 | 18/28 | 22/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=26) | 4, 8 and 12mg Tirzepatide (N=29) | 2.5, 5, 10, and 15mg Tirzepatide (N=28) | 2.5, 7.5 and 15mg Tirzepatide (N=28)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=26) | 4, 8 and 12mg Tirzepatide (N=29) | 2.5, 5, 10, and 15mg Tirzepatide (N=28) | 2.5, 7.5 and 15mg Tirzepatide (N=28)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (9) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 5 (5) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (2) | 2 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (5) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 9 (18) | 10 (19) | 9 (19)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 5 (7) | 3 (12) | 3 (3)
Eructation (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 2 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 7 (14) | 11 (18) | 10 (16)
Vomiting (Gastrointestinal disorders) | 1 (1) | 5 (6) | 5 (7) | 5 (7)
Fatigue (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 2 (3) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 6 (7) | 8 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (9)
Headache (Nervous system disorders) | 2 (2) | 2 (5) | 6 (10) | 5 (27)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 2 (2) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-08-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT03311724/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT03311724/SAP_001.pdf